CLINICAL TRIAL: NCT05517785
Title: The Effect of Pharmacological Treatment for ADHD on Physical Performance in Male Adolescents
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Loewenstein Hospital (Other)
Collaborators: Wingate Institute (Other)
Responsible Party: Principal Investigator, Aviva Mimouni-Bloch, Head of Child Developmental Center, Loewenstein Hospital
Other Study IDs: 0003-22-LOE
Record Dates: First submitted 2022-08-16; First posted 2022-08-26 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Medicated: Assessment of motor function will be performed 1 hour after taking the usual stimulant ADHD medication.
  Interventions: Other: Motor performance tests
- Unmedicated: Participants will remain unmedicated for the duration of the assessment, and will delay taking their usual stimulant ADHD medication until all the motor function assessments are completed.
  Interventions: Other: Motor performance tests

INTERVENTIONS:
Other: Motor performance tests — Performance of 5 motor tests: plank, single leg stance test, standing long jump test (broad jump), 4 x 10 agility test and 20 m shuttle run tests (beeps), after taking ADHD drug or not taking the drug before motor tests performance

SUMMARY:
The aim of this study is to evaluate the effects of stimulant ADHD pharmacotherapy on motor performance in male adolescents.

DETAILED DESCRIPTION:
This study is designed as a single-center, crossover, randomized study. 70 high-school aged males aged between 15 and 18 years with a diagnosis of ADHD who are being treated pharmacologically using stimulants (such as Ritalin, Concerta, Vyvanse etc) will be recruited. The study will investigate motor performance using several motor function tests both with and without the influence of stimulant ADHD medications.

Participants will be assessed on two separate occasions, both sessions will occur during the morning in their regular school environment. During the sessions, participants will be randomized, 50% will be assessed one hour after taking their usual stimulant ADHD medication and the other 50% will be asked to postpone taking their usual stimulant ADHD medication until the session is finished. During the two separate sessions, all participants will be asked to perform the following motor tests: plank, single leg stance test, standing long jump test (broad jump), 4 x 10 agility tests and 20 m shuttle run tests (beeps).

ELIGIBILITY:
Inclusion Criteria:

* High school male students
* Diagnosis of ADHD
* Treatment with prescribed stimulants for ADHD (e.g. Concerta, Ritalin, Phenidin, Focalin etc.).

Exclusion Criteria:

* Students with concomitant chronic disease (including asthma, cardiac, motor, neurological and gastrointestinal disturbances)
* History of acute illness in the previous two weeks
* Any injuries that would inhibit the ability to exercise or play sport
* Students unable to obtain parental/guardian consent
* Students unwilling to participate

Ages: 15 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — This research will analyze physiological data that is sex dependent
Study Population: 70 high school boys ages 15-18 years, diagnosed with ADHD and treated with stimulant medications
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Motor tests | 5 minutes
  Plank
Motor tests | 5 minutes
  Single leg stance test
Motor tests | 5 minutes
  Standing long jump test (broad jump)
Motor tests | 5 minutes
  4 x 10 agility tests
Motor tests | 5 minutes
  20 m shuttle run tests (beeps)
AAC-Q questionnaire | 10 minutes
  Adolescents and Adults Coordination Questionnaire

SECONDARY OUTCOMES:
Heart rate at rest | 5 minutes
  Heart rate will be measured in a sitting position
Blood pressure at rest | 5 minutes
  Blood pressure will be measured in a sitting position

CONTACTS AND LOCATIONS:
Locations (1):
- Sharon Tsuk, Netanya, Israel

IPD SHARING:
Plan to Share IPD: Undecided